CLINICAL TRIAL: NCT06142201
Title: A Real-world Study：Disease Outcome and Safety of JT001 in Patients With Coronavirus Disease 2019 (COVID-19)
Brief Title: A Real-World Study of JT001 for COVID-19
Status: Active, not recruiting | Type: Observational
Sponsor: Shanghai Vinnerna Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: JT001-PMS-CO02-COVID-19
Record Dates: First submitted 2023-11-20; First posted 2023-11-21 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — GS-621763

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- JT001
  Interventions: Drug: JT001
- No anti-SARS-CoV-2 treatment
  Interventions: Drug: JT001

INTERVENTIONS:
Drug: JT001 — oral administration
  Other Names: DeuremidevirHydrobromideTablets

SUMMARY:
Real-world disease outcomes and safety in patients with mild to moderate COVID-19 treated with JT001

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old.
2. The novel coronavirus infection (COVID-19) meets at least one of the following five criteria:

1) Diagnosis of novel coronavirus infection; 2) Diagnosed with novel coronavirus pneumonia; 3) The novel coronavirus nucleic acid test is positive; 4) Test positive for novel coronavirus antigen; 5) Culture positive for novel coronavirus.

3. Patients who have not developed severe COVID-19 or died within 28 days of COVID-19 diagnosis, or who have developed severe COVID-19 or died within 28 days of COVID-19 diagnosis, were treated with deuterimodivir hydrobromide tablets or were not treated with anti-novel coronavirus before disease progression.

Exclusion Criteria:

· Patients who have not developed severe COVID-19 or died within 28 days of COVID-19 diagnosis, or those who have developed severe COVID-19 or died within 28 days of COVID-19 diagnosis, received the following anti-novel coronavirus treatments before disease progression, including: Nematavir tablet/Ritonavir tablet, Azvudine tablet, Monoravir capsule, Zenotavir tablet/Ritonavir tablet, Leritvir tablet, Ambavirzumab/Romisivir injection, human immunoglobulin for COVID-19 or convalescent plasma for COVID-19 survivors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with mild to moderate COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 7656 (Actual)
Dates: Start 2023-08-31 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of COVID-19 disease progression (severe COVID-19 or all-cause death) by day 28 | Within 28 days
  Incidence of COVID-19 disease progression (severe COVID-19 or death from any cause) at day 28 from COVID-19 diagnosis. According to the diagnosis of severe COVID-19 and indicators meeting the diagnostic definition of severe COVID-19, the evaluation and analysis were performed.

SECONDARY OUTCOMES:
Incidence of the following COVID-19 disease progression events by day 28 | Within 28 days
  Severe COVID-19 or all-cause death in patients with high-risk factors,Elderly patients (≥65 years) with severe COVID-19 or all-cause death,All enrolled patients had severe COVID-19,All enrolled patients died from all causes,COVID-19 related hospitalizations in non-hospitalized patients,Hospitalized patients with severe COVID-19 or all-cause death.
Incidence of severe Covid-19-related events up to day 28 | Within 28 days
  Incidence of severe Covid-19-related events up to day 28,Respiratory rate ≥30 times/min, Oxygen saturation (SpO2) ≤93% ,Partial oxygen pressure (PaO2)/Oxygen concentration (FiO2) ≤300mmHg,Lung imaging showed significant lesion progression > 50% within 24 to 48 hours,Mechanical ventilation o Respiratory failure and mechanical ventilation,Shock,Stay in ICU,Organ failure and admission to ICU.
The incidence of all aes and abnormal laboratory changes on day 28, etc | Within 28 days
  The incidence of all aes and abnormal laboratory changes on day 28, etc

OTHER OUTCOMES:
Changes of SARS-CoV-2 through Day 28 | Within 28 days
  Percentage of patients who achieve SARS-CoV-2 nucleic acid negative through Day 28，Change of SARS-CoV-2 viral load from baseline to Day 28

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - Peking university first hospital, Beijing, Beijing Municipality
  - Shanghai Fourth People's Hospital, Shanghai, Shanghai Municipality
  - Longhua Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality
  - Gongli Hospital, Pudong New Area, Shanghai, Shanghai, Shanghai Municipality
  - Central Hospital of Minhang District, Shanghai, Shanghai, Shanghai Municipality
  - Shanghai Pudong Hospital, Fudan University Affiliated Pudong Medical Center, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No